CLINICAL TRIAL: NCT04784351
Title: Prediction of Expected Length of Hospital Stay Using Machine Learning
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Biofourmis Inc. (Industry)
Responsible Party: Principal Investigator, David Levine, Attending Physician, Brigham and Women's Hospital
Other Study IDs: 2017P002583b
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Infection; Heart Failure; Chronic Obstructive Pulmonary Disease; Asthma; Gout Flare; Chronic Kidney Diseases; Hypertensive Urgency; Atrial Fibrillation Rapid; Anticoagulants; Increased
MeSH Terms: conditions — Infections; Heart Failure; Pulmonary Disease, Chronic Obstructive; Asthma; Renal Insufficiency, Chronic; Hypertensive Crisis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training: A subset of patients that are used to train the machine learning algorithm.
- Validation: A subset of patients that are "held back" and used to validate the algorithm's accuracy.

SUMMARY:
This is a retrospective observational study drawing on data from the Brigham and Women's Home Hospital database. Sociodemographic and clinic data from a training cohort were used to train a machine learning algorithm to predict length of stay throughout a patient's admission. This algorithm was then validated in a validation cohort.

ELIGIBILITY:
Was a subject in the Brigham and Women's Home Hospital study and has a completed record in the study's database.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted at Brigham and Women's Hospital and Brigham and Women's Faulkner Hospital who meet primary diagnosis, age, and residence within 5 mile requirements and are enrolled in home hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-03-20 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Length of Stay | From date of admission to date of discharge (1 to 24 days)
  The time spent by each patient in Home Hospital from time of admission to time of discharge, measured in hours

CONTACTS AND LOCATIONS:
Overall Officials: David Levine, MD MPH MA, Principal Investigator — Associate Physician
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lubelski D, Ehresman J, Feghali J, Tanenbaum J, Bydon A, Theodore N, Witham T, Sciubba DM. Prediction calculator for nonroutine discharge and length of stay after spine surgery. Spine J. 2020 Jul;20(7):1154-1158. doi: 10.1016/j.spinee.2020.02.022. Epub 2020 Mar 13. PMID 32179154
- [Background] Karnuta JM, Churchill JL, Haeberle HS, Nwachukwu BU, Taylor SA, Ricchetti ET, Ramkumar PN. The value of artificial neural networks for predicting length of stay, discharge disposition, and inpatient costs after anatomic and reverse shoulder arthroplasty. J Shoulder Elbow Surg. 2020 Nov;29(11):2385-2394. doi: 10.1016/j.jse.2020.04.009. Epub 2020 Jun 9. PMID 32713541
- [Background] Ramkumar PN, Navarro SM, Haeberle HS, Karnuta JM, Mont MA, Iannotti JP, Patterson BM, Krebs VE. Development and Validation of a Machine Learning Algorithm After Primary Total Hip Arthroplasty: Applications to Length of Stay and Payment Models. J Arthroplasty. 2019 Apr;34(4):632-637. doi: 10.1016/j.arth.2018.12.030. Epub 2018 Dec 27. PMID 30665831
- [Background] Ma X, Si Y, Wang Z, Wang Y. Length of stay prediction for ICU patients using individualized single classification algorithm. Comput Methods Programs Biomed. 2020 Apr;186:105224. doi: 10.1016/j.cmpb.2019.105224. Epub 2019 Nov 20. PMID 31765937
- [Background] Daghistani TA, Elshawi R, Sakr S, Ahmed AM, Al-Thwayee A, Al-Mallah MH. Predictors of in-hospital length of stay among cardiac patients: A machine learning approach. Int J Cardiol. 2019 Aug 1;288:140-147. doi: 10.1016/j.ijcard.2019.01.046. Epub 2019 Jan 19. PMID 30685103
- [Background] Bacchi S, Oakden-Rayner L, Menon DK, Jannes J, Kleinig T, Koblar S. Stroke prognostication for discharge planning with machine learning: A derivation study. J Clin Neurosci. 2020 Sep;79:100-103. doi: 10.1016/j.jocn.2020.07.046. Epub 2020 Aug 5. PMID 33070874
- [Background] Navarro SM, Wang EY, Haeberle HS, Mont MA, Krebs VE, Patterson BM, Ramkumar PN. Machine Learning and Primary Total Knee Arthroplasty: Patient Forecasting for a Patient-Specific Payment Model. J Arthroplasty. 2018 Dec;33(12):3617-3623. doi: 10.1016/j.arth.2018.08.028. Epub 2018 Sep 5. PMID 30243882
- [Background] Young AJ, Hare A, Subramanian M, Weaver JL, Kaufman E, Sims C. Using Machine Learning to Make Predictions in Patients Who Fall. J Surg Res. 2021 Jan;257:118-127. doi: 10.1016/j.jss.2020.07.047. Epub 2020 Aug 18. PMID 32823009
- [Background] Sinha I, Aluthge DP, Chen ES, Sarkar IN, Ahn SH. Machine Learning Offers Exciting Potential for Predicting Postprocedural Outcomes: A Framework for Developing Random Forest Models in IR. J Vasc Interv Radiol. 2020 Jun;31(6):1018-1024.e4. doi: 10.1016/j.jvir.2019.11.030. Epub 2020 May 4. PMID 32376173
- [Background] Merrill RK, Ferrandino RM, Hoffman R, Shaffer GW, Ndu A. Machine Learning Accurately Predicts Short-Term Outcomes Following Open Reduction and Internal Fixation of Ankle Fractures. J Foot Ankle Surg. 2019 May;58(3):410-416. doi: 10.1053/j.jfas.2018.09.004. Epub 2019 Feb 23. PMID 30803914
- [Background] Nemati M, Ansary J, Nemati N. Machine-Learning Approaches in COVID-19 Survival Analysis and Discharge-Time Likelihood Prediction Using Clinical Data. Patterns (N Y). 2020 Aug 14;1(5):100074. doi: 10.1016/j.patter.2020.100074. Epub 2020 Jul 4. PMID 32835314